CLINICAL TRIAL: NCT04806841
Title: Effect of a Motivational Intervention on Exercise Adherence After Cardiac Rehabilitation
Acronym: IMREADAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Bherer (Other)
Responsible Party: Sponsor-Investigator, Louis Bherer, Associate scientific director, Direction of prevention, Montreal Heart Institute, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-2235
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2021-06

CONDITIONS: Aging
Keywords: Aging; Motivation; Cardiac rehabilitation; Exercise adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants will have access to 4 weekly supervised training sessions for 3 months. The intervention group will also take part in 3 group meetings (behavioral intervention) and will receive follow-up phone calls from month 4 to 6.
  Interventions: Behavioral: Motivational intervention
- Control group (Experimental): Participants will have access to 4 weekly supervised training sessions for 3 months without any behavioral intervention.
  Interventions: Other: Control intervention

INTERVENTIONS:
Behavioral: Motivational intervention — Three group meeting of 60 minutes to help create effective goals and methods on maintaining motivation to exercise regularly. These meetings will help participants create effective goals and methods on maintaining their motivation to exercise regularly. They will then receive a monthly phone call follow-up at months 4-6.
  Arms: Intervention group
Other: Control intervention — Participants in the control group will be simply encouraged to exercise at the EPIC center and complete the online surveys. Participants in the control group will receive the skills/tactics at the end of the study.
  Arms: Control group

SUMMARY:
The Canadian Physical Activity Guidelines recommend that adults should exercise for at least 150 minutes per week. Incorporating 150 minutes of moderate-to-vigorous intensity physical activity (MVPA) a week has been associated with the prevention of at least 25 chronic diseases, including cardiovascular disease. However, most people do not successfully maintain this active behavior. The primary objective of this investigation is to understand what predicts successful exercise adherence and why people dropout from the gym. The long-term impact of this study has implications for future policy level interventions aimed at exercise adherence.

DETAILED DESCRIPTION:
The participants will receive a link to the baseline survey at www.surveymonkey.com. After completing the survey, the participants will be randomized into an intervention or a control group. The intervention group will be invited to attend a group meeting at weeks 1, 6 and 12 (3-month mark) which will take place at the EPIC center. These meetings will help participants create effective goals and methods on maintaining their motivation to exercise regularly. The participants will then receive a monthly phone call follow-up at months 4-6. The purpose of these meeting/follow-ups is to serve as a review of the worksheet, address any questions and help make any modification plans if necessary. Participants in the control group will be simply encouraged to exercise at the EPIC center and complete the online surveys. Participants in the control group will receive the skills/tactics at the end of the study. As members of the EPIC center, all participants will have access to four weekly supervised sesssions for three months.

ELIGIBILITY:
Inclusion Criteria:

* 50 years and older, included in the prevention clinique at Epic Center after an acute coronary syndrome (≤ 12 months) with or without revascularization, doing less than 150 minutes of physical activity per week. The approval of a cardiologist is needed to take part in this program. A normal score on the MoCA (≥ 26) is needed.

Exclusion Criteria:

* Valve surgery without any coronary event, non-cardiopulmonary exercise limitation, stress induce malignant arrhythmia and decompensate heart failure

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Physical activity level | Baseline and 6 months
  Godin Leisure Time Exercise Questionnaire (GLTEQ). Frequency and duration are open-ended questions with 0 set as minimum and with no maximum. Higher value indicates greater participation in physical activity.

SECONDARY OUTCOMES:
Behavioral automaticity | Baseline and 6 months
  Self-Report Behavioral Automaticity Index (SRBAI) The complete name of the scale is the "Self-Report Behavioral Automaticity Index". The scores on this scale range from 1 to 5, with 1 indicating less use of automatic process and 5 indicating a strong use of automatic processes when exercising. Higher scores are preferrable/represent better outcome as they indicate that exercise behavior is performed easily.
Autoregulation / Self-control | Baseline and 6 months
  Self-reported activity journal
Behavioral regulation | Baseline and 6 months
  Intrinsic regulation subscale from the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2). Behavioral Regulation was assessed by a scale proposed by Sniehotta, Scholz, & Schwarzer (2006), which does not have a specific title. The scores on this scale range from 1 to 5, with 1 indicating less use of planning and 5 indicating a strong use of planning for their exercise sessions. Higher scores are preferrable/represent better outcome as they indicate that participants make plans to schedule their exercise sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bherer, PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Preventive medicine and physical activity centre (centre EPIC), Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhodes RE, de Bruijn GJ. What predicts intention-behavior discordance? A review of the action control framework. Exerc Sport Sci Rev. 2013 Oct;41(4):201-7. doi: 10.1097/JES.0b013e3182a4e6ed. PMID 23873134
- [Background] Kaushal N, Rhodes RE. Exercise habit formation in new gym members: a longitudinal study. J Behav Med. 2015 Aug;38(4):652-63. doi: 10.1007/s10865-015-9640-7. Epub 2015 Apr 8. PMID 25851609
- [Background] Kaushal N, Rhodes RE, Spence JC, Meldrum JT. Increasing Physical Activity Through Principles of Habit Formation in New Gym Members: a Randomized Controlled Trial. Ann Behav Med. 2017 Aug;51(4):578-586. doi: 10.1007/s12160-017-9881-5. PMID 28188586
- [Background] Warburton DE, Katzmarzyk PT, Rhodes RE, Shephard RJ. Evidence-informed physical activity guidelines for Canadian adults. Can J Public Health. 2007;98 Suppl 2:S16-68. PMID 18213940
- [Background] Blanchard CM. Heart disease and physical activity: looking beyond patient characteristics. Exerc Sport Sci Rev. 2012 Jan;40(1):30-6. doi: 10.1097/JES.0b013e318234c206. PMID 21918456
- [Background] Schulz KF, Grimes DA. Sample size calculations in randomised trials: mandatory and mystical. Lancet. 2005 Apr 9-15;365(9467):1348-53. doi: 10.1016/S0140-6736(05)61034-3. PMID 15823387
- [Background] Godin G, Jobin J, Bouillon J. Assessment of leisure time exercise behavior by self-report: a concurrent validity study. Can J Public Health. 1986 Sep-Oct;77(5):359-62. No abstract available. PMID 3791117
- [Background] Godin G, Shephard RJ, Colantonio A. The cognitive profile of those who intend to exercise but do not. Public Health Rep. 1986 Sep-Oct;101(5):521-6. PMID 3094084
- [Background] Gardner B, Abraham C, Lally P, de Bruijn GJ. Towards parsimony in habit measurement: testing the convergent and predictive validity of an automaticity subscale of the Self-Report Habit Index. Int J Behav Nutr Phys Act. 2012 Aug 30;9:102. doi: 10.1186/1479-5868-9-102. PMID 22935297
- [Background] Carver CS, Scheier MF. Control theory: a useful conceptual framework for personality-social, clinical, and health psychology. Psychol Bull. 1982 Jul;92(1):111-35. No abstract available. PMID 7134324
- [Background] Shek DT, Ma CM. Longitudinal data analyses using linear mixed models in SPSS: concepts, procedures and illustrations. ScientificWorldJournal. 2011 Jan 5;11:42-76. doi: 10.1100/tsw.2011.2. PMID 21218263
- [Background] West BT. Analyzing longitudinal data with the linear mixed models procedure in SPSS. Eval Health Prof. 2009 Sep;32(3):207-28. doi: 10.1177/0163278709338554. Epub 2009 Aug 13. PMID 19679634